CLINICAL TRIAL: NCT00557050
Title: Acute Hamstring Strains in Danish Elite Soccer - Prevention and Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Amager Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-A-2007-0062
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2007-11-12 (Estimated); Status verified 2007-09

CONDITIONS: Strains
Keywords: Hamstring; Muscle; Injury; Prevention; Muscles
MeSH Terms: conditions — Sprains and Strains; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Training — 10-week eccentric hamstring muscle training

SUMMARY:
A common soft tissue injury in sports involving sprinting and jumping is the hamstring strain.

Not much evidence-based research has been carried out on prevention of hamstring strains.

Most studies suggest that hamstring strains occur during the later part of the swing phase when the player is sprinting. In this phase the hamstring muscles are working to decelerate knee extension - that is, the muscle develops tension while lengthening. This means that the muscles change from functioning eccentrically to concentrically. We hypothesize that it is during this rapid change from eccentric to concentric function that the muscles are most vulnerable to injuries, and that the injuries can be prevented by increasing the eccentric muscle strength in the hamstring.

This randomized clinical trial will examine the effect of a 10-week preseason strength-training program in Danish elite soccer. The strength-training program focuses on eccentric hamstring training.

60 elite teams (1200 soccer players) will be cluster-randomized to either ordinary training or ordinary training combined with eccentric hamstring strength training. The training group will start the training program in the pre-season (10 weeks) and continue the training once a week during the following season.

Suspected hamstrings strains during the season will be examined within 3 days using ultrasound. Ultrasound verified hamstring strains will be registered, and players will start a standardized rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Male soccer player in one of the top 4 divisions i Denmark in the 2007/08 season
* Minimum 18 years old at the time for inclusion

Exclusion Criteria:

* Current hamstring strain at the time for inclusion
* Under 18 years old

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2008-01; Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Number of acute hamstring strains | one soccer season

SECONDARY OUTCOMES:
Number of ACL-injuries | One soccer season

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Petersen, MD, Principal Investigator — Department of Orthopaedic Surgery, Amager University Hospital, Denmark

REFERENCES:
- [Background] Petersen J, Holmich P. Evidence based prevention of hamstring injuries in sport. Br J Sports Med. 2005 Jun;39(6):319-23. doi: 10.1136/bjsm.2005.018549. PMID 15911599